CLINICAL TRIAL: NCT03447158
Title: Effects of Hyperosmolar Dextrose Injection in Rotator Cuff Disorder With Bursitis : A Randomized Controlled Trial
Brief Title: Effects of Hyperosmolar Dextrose in Rotator Cuff Disorder With Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18MMHIS001
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Subacromial Bursitis
MeSH Terms: interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15% Dextrose group (Experimental): 4.5cc 15% dextrose and 0.5cc 1% xylocaine was injected into inflamed subacromial bursa under sonographically guidance
  Interventions: Procedure: 15% Dextrose
- control group (Placebo Comparator): 4.5cc normal saline and 0.5cc 1% xylocaine was injected into inflamed subacromial bursa under sonographically guidance
  Interventions: Procedure: Normal saline

INTERVENTIONS:
Procedure: 15% Dextrose — inject 15% dextrose and xylocaine into subacrominal bursa under sonographically guidance
  Arms: 15% Dextrose group
Procedure: Normal saline — inject normal saline and xylocaine into subacrominal bursa under sonographically guidance
  Arms: control group

SUMMARY:
The main purpose of this study is to compare treatment efficacy of different concentration dextrose injection in chronic subacromial bursitis .

DETAILED DESCRIPTION:
Rotator cuff disorder with bursitis is one of the most frequent pathologies of the shoulder, which may cause serious restriction of daily activities and reduce quality of life. There are many ways in treating rotator cuff disorder with bursitis, including medication, physical therapy, kinesiological taping, acupuncture and local injection. Protholotherapy, which inject hyperosmolar dextrose to soft tissue, is a novel management in musculoskeletal disorders. However, only few trials exist in studying hyperosmolar dextrose injection for rotator cuff disorder with bursitis and most of them have small sample size and not randomized. The aim of this study was to figure out the effects of sonographically guided subacromial bursa injection with hyperosmolar dextrose in rotator cuff disorder with bursitis by a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. 20-65 years-old
2. pain lasting >3 months
3. Painful arc between 40° to 120° in abduction
4. positive Neer and Hawkins-Kennedy tests
5. positive Empty can test
6. pain in daily living activities
7. Bursa thickness more than 2mm in ultrasound
8. Rotator cuff tendinopathy

Exclusion Criteria:

1. history of significant shoulder trauma
2. history of surgery, fracture, or dislocation
3. adhesive capsulitis
4. full thickness rotator cuff tear
5. a long head of bicep tendon tear
6. Contra-indications to local dextrose injection (known blood coagulation disorders, warfarin therapy, allergy to dextrose)
7. previous shoulder steroid injection in one month
8. had any rheumatologic, systemic, or neurologic disorders
9. patients taking regular systemic NSAIDs or steroids
10. pregnant or breastfeeding mothers
11. malignancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline pain on activity at 1 week, 1 month, and 3 months after 3rd section of therapy | before therapy sections, 1 week, 1 month, and 3 months after 3rd section of therapy
  maximal visual analog scale (VAS) in the past week during shoulder activity. Visual analog scale is range from 0-10. The higher score indicated more severe pain.

SECONDARY OUTCOMES:
Change from Baseline shoulder joint active range of motion (PROM) at 1 week, 1 month, and 3 months after 3rd section of therapy | before therapy sections, 1 week, 1 month, and 3 months after 3rd section of therapy
  abduction and flexion
Change from Baseline Shoulder Pain and Disability Index (SPADI) score at 1 week, 1 month, and 3 months after 3rd section of therapy | before therapy sections, 1 week, 1 month, and 3 months after 3rd section of therapy
  Shoulder pain and disability questionnaire with two subscales, pain scale and function scale. Pain scale is range from 0-50. The higher scale indicates worse pain outcome. Function scale is range from 0-80. The higher scale indicates poor shoulder function. The total scale is summation of pain scale and function scale.
Change from Baseline Ultrasound property at 1 week, 1 month, and 3 months after 3rd section of therapy | before therapy sections, 1 week, 1 month, and 3 months after 3rd section of therapy
  Thickness of bursa and elastogram
Change from Baseline pain on resting at 1 week, 1 month, and 3 months after 3rd section of therapy | before therapy sections, 1 week, 1 month, and 3 months after 3rd section of therapy
  maximal visual analog scale (VAS) in the past week during resting. Visual analog scale is range from 0-10. The higher score indicated more severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang YJ, Chang FH, Hou PH, Tseng KH, Lin YN. Effects of Hyperosmolar Dextrose Injection in Patients With Rotator Cuff Disease and Bursitis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Feb;102(2):245-250. doi: 10.1016/j.apmr.2020.08.010. Epub 2020 Sep 11. PMID 32926850